CLINICAL TRIAL: NCT04488432
Title: Endocrine, Bone And Metabolic Disorders In Adults After Allogeneic Stem-cell Transplant
Acronym: ENDOCALLOGREFF
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0137
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Endocrine System Diseases; Osteoporosis; Metabolic Syndrome; Adrenal Insufficiency
MeSH Terms: conditions — Endocrine System Diseases; Osteoporosis; Metabolic Syndrome; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Allogeneic hematopoietic stem cell transplantations (allo-HSCT) is often indicated in malignant hematologic diseases. Conditioning regimens, used to reduce the tumor burden and to prevent transplant rejection, are based on chemotherapy alone or combined with total body irradiation (TBI). Endocrine complications are frequent transplant-related side effects. Investigators have been well described in children studies but less in adulthood.

The objective of this study is to assess retrospectively endocrine, bone and metabolic disorders in adult patients, 12 months after allo-HSCT.

DETAILED DESCRIPTION:
Patients & Methods Inclusion criteria are : patients treated with allo-HSCT from 2006 to 2016 for a malignant hematologic disease; adult and in complete remission at exploration.

Exclusion criteria are : anteriority of brain radiotherapy and prior HSCT.

Twelve months after HSCT, each patient underwent fasting measurement of IGF1, TSH, fT4, FSH, LH, sex steroids, glycemia, insulin level, and lipid profile. Unless contraindication, adrenal and growth hormone functions were assessed with insulin hypoglycemia test. A dual X-ray absorptiometry was also performed.

Investigators will assess the prevalence of endocrine, bone and metabolic disorders 12 months after allo-HSCT and describe some of their risk factors.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with allo-HSCT from 2006 to 2016 for a malignant hematologic disease
* adult and in complete remission at exploration.

Exclusion Criteria:

* anteriority of brain radiotherapy
* prior HSCT
* pregnancy

Ages: 16 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with allo-HSCT after puberty from 2006 to 2016 in our University Hospital of Brest, adult at the endocrine exploration.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Adrenal insuffisiency prevalence | 12 month post-alloHSCT
  insulin hypoglycemia test

SECONDARY OUTCOMES:
Hypothyroidism prevalence | 12 month post-alloHSCT
  fT4, TSH
Growth hormon Deficiency prevalence | 12 month post-alloHSCT
  insulin hypoglycemia test
Premature ovarian failure prevalence | 12 month post-alloHSCT
  FSH, LH, estradiol
Prevalence of elevated FSH in men | 12 month post-alloHSCT
  FSH, testosterone
Prevalence of low bone mineral density | 12 month post-alloHSCT
  dual X-ray absorptiometry
Prevalence of obesity | 12 month post-alloHSCT
  BMI
Prevalence of dyslipidemia | 12 month post-alloHSCT
Prevalence of hyperglycemia and insulin-resistance | 12 month post-alloHSCT
  glycemia and HOMA2-IR index

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest - Endocrinology and Diabetology Department, Brest, France

IPD SHARING:
Plan to Share IPD: No